CLINICAL TRIAL: NCT04313738
Title: Effects of Home-Based Nursing Interventions Performed in Accordance With The Transtheoretical Model on Smoking Cessation in Patients With The Chronic Obstructive Pulmonary Disease: Randomised Controlled Trial
Brief Title: Transtheoretical Model Based Nursing Interventions on Smoking Cessation in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Figen Cavusoglu, Assistant Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ODM.0.20.08/1184
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: COPD; Smoking Cessation; Home Visit
Keywords: COPD; Smoking cessation; Transtheoretical model; Home visit; Nursing; Motivational interview
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Masking Description: The study had a single-blind, randomized controlled experimental design. To avoid bias, participants were not told whether they were in the experimental or the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Experimental: Intervention group Intervention group: Home visit, health education, telephone counseling At the intervention group; the researcher firstly made spirometry meausurement in hospital. After, the researcher made pretest (baseline measurement) before nursing interventions at the first home visit. At the first home visit, the researcher was offered education and guide smoking cessation. Second, Third and fourth home visit were made 15 days later, one and six months after visit first visit. During the second, third and fourth home visits, firstly the patient's stage of change was determined and then appropriate nursing intervention was performed in accordance with the guidelines.Between the third and fourth home visits, the participants were contacted through telephone calls once a month. At fourth home visit, the researcher made posttest. After the patient was invited to the hospital and spirometry measurements were repeated.
  Interventions: Other: Assigned Interventions
- Control Group (No Intervention): At the control group; No home visits were paid to the control group. The researcher made measurements twice at in the first and sixth months in the hospital. The researcher also given at the end of the sixth month, all of the nursing interventions, given to the intervention group, for the control group.

INTERVENTIONS:
Other: Assigned Interventions — Home visit, health education
  Arms: Intervention group

SUMMARY:
Background: The aim of this study is to evaluate the efficiency of nursing intervention based on smoking cessation transtheoretical model in patients with COPD who smoke Method: Experimental design was used in the study. Thirty-three patients in the study group were completed with 35 chronic obstructive pulmonary disease patients in the control group. Sociodemographic characteristics data form, Fagerstrom Nicotine Dependency Test, Transteoretic Model Decision Making Scale, Self-efficacy Scale, Change Stages Scale and Behavior Modification Scale were used as data collection form. In the analysis of the data, the significance test of the difference between the two means, the significance test of the difference between two peers, the two-ratio test, Chi square, Mann Withney U test and Wilcoxon test were used.

Results: Decision-making subscale scores, self-efficacy score scores, and behavior modification methods subscale scores showed significant increases (p<.05) in the decision-making subscale of the patients in the experimental group after the home nursing interventions (p<.05). While there was a significant improvement in the change stages, 9 patients in the experimental group and 2 patients in the control group had left the cigarette but the difference between them was significant (p<.05).

What does this paper contribute?

* Nursing interventions with home visits based on transtheoretical model supplied to quit smoking of patients
* The nursing interventions with home visits based on transtheoretical model contributed positively to behavioral change in patients' smoking cessation.

DETAILED DESCRIPTION:
Aim of the study The present study was aimed at investigating the effects of nursing interventions on the outcomes of smoking cessation in patients with COPD who smoke.

Study design and setting The study had a single-blind, randomized controlled experimental design. To avoid bias, the participants were not told whether they were in the experimental or the control group. The conceptual structure of the study is given in Figure 1. This randomized clinical trial was based on the guidelines proposed by the Consolidated Standart of Reporting Trials-CONSORT 2010 (Supplementary file 1). The study was conducted between January 2016 and November 2017 at hospital and at homes of the patients with COPD enrolled in a public special branch hospital

Randomization An intervention group and a control group formed by using the research randomizer software. The program used random numbers to select participants and randomly assign them to the experimental or control group (600 participants were assigned to each group). Homogeneity test showed no significant difference between the measures of the groups in table 1 (p>.05).

Blinding of data collectors and the statistician was implemented in this randomized blinded study. Another researcher who did not know the group assignments coded the data in the computer. After statistical analysis was conducted and research report was written, asisstant researcher explained the codes for experimental and control group. Therefore, blinding of the collectors, statistical analysis, and report writing was provided.

Study outcomes, The tools used to collect the data were as follows: Sosyodemographic characteristics questionnaire, Fagerström Test for Nicotine Dependence (FTND) and the components of the Transtheoretical model (Stages of Change (SOC) scale, Processes of Change (POC) scale, Self-Efficacy (SE) scale and Decisional Balance (DB) scale. In addition, measurements were performed using the spirometry available in the hospital where data were collected.

Fagerström Test for Nicotine Dependence: The test includes 6 items each of which is rated on a different scale. A total score ranging from 0 to 4 indicates low nicotine dependence, from 5 to 6 indicates moderate dependence and from 7 to 10 indicates high independence. The validity and reliability study of the Turkish version of the scale was conducted. While the coefficient alpha value of the original scale was 0.61, cronbach's alpha value was 0.56 in Turkish version' validity and reliability study and 0.79 in the present study.

Stages of Change (SOC) scale: Prochaska and Diclemente (1983) explained smoking cessation through the gradual change process and developed the questions of change. Accordingly, people select one of the following corresponding to his/her situation: Precontemplation: I do not consider quitting smoking in the next six months. Contemplation: I am planning to quit smoking in the next six months. Preparation: I am planning to quit in the next 30 days. Action: I quit smoking less than six months ago. Maintenance: I have not been smoking for more than six months.

Processes of Change (POC) scale: The scale includes 30 items questioning the cognitive processes (15 items) and behavioral processes (15 items). Each process contains five sub-dimensions. It is a five-point Likert type scale ranging from 1 to 5 (1=never, 2=rarely, 3=occasionally, 4=often, 5=very often). The options determine which methods an individual uses in behavior change. Coefficient Alpha values range between 0.78 and 0.91. Cronbach's Alpha values of the Turkish version of the scale whose validity and reliability study was conducted ranged between 0.54 and 0.86. In the present study, Cronbach's Alpha values ranged between 0.61 and 0.92.

Self-Efficacy (SE) scale: The scale measures the degree of confidence an individual has in maintaining non-smoking behavior in situations triggering smoking. The validity and reliability study of the Turkish version of the scale was conducted. While the coefficient alpha value of the original scale was 0.82, Cronbach's alpha values of was 0.85 in Turkish version's validity and reliability study and 0.93 in the present study. The scale consists of eight items rated on a 5-point Likert type scale ranging from 1 to 5 (1=not confident at all, 2=a little confident, 3=confident, 4=very confident and 5=extremely confident). The lowest and highest possible scores to be obtained from the scale are 8 and 40 respectively. The higher the score is the more successful the person is.

Decisional Balance (DB) scale: The scale has 12 items in two sub-dimensions: Pros of change (6 items) and Cons of change (6 items). The Coefficient Alpha value used to calculate the internal validity of the original scale and was 0.87for the Pros of change subscale and 0.90 for the Cons of change subscale.

The Cronbach's Alpha value for the Pros of change and Cons of change subscales was 0.88 and 0.82 in the Turkish version' and 0.71 and 0.85 in the present study. The items of the scale are rated on a five-point likert type scale ranging from 1 to 5 (1=not important at all, 2=very little important, 3=moderately important, 4=very important and 5=extremely important). The minimum and maximum possible scores to be obtained from the scale are 6 and 30 respectively. While high Pros of change subscale scores indicate that the individual is determined to change, high Cons of change subscale scores indicate that the person is not aware of the harms of the problematic behavior.

Study protocol Oral informed consent was obtained from eligible patients with COPD at initial interviews on the phone. The patients with COPD who agreed to participate in the study were assigned to the groups according to the research randomizer software. The patients in the intervention group and the control group separately were first invited to the hospital and obtain written informed consent was obtained at first interview.

At the intervention group; The researcher made spirometry measurements in the hospital. then appointment were made for the first of the four planned visits. In the first home visit, the aim and the process of the project were explained, the patient's stage of change was determined by administering the scales, and a TTM-based nursing intervention related to smoking cessation and COPD management was applied. The nursing intervention performed in the present study involved home visits and six-month periodic follow-up, health education, smoking cessation intervention in line with motivational interviewing principles and telephone counseling processes. During the second, third and fourth home visits, first, the patient's stage of change was determined and then appropriate nursing intervention was performed in accordance with the guidelines. Given his/her needs, the patient was informed about the disease using the training booklet and the booklet was given to the patient. Between the third and fourth home visits, the participants were contacted through telephone calls once a month to ensure the continuity of the motivation and thus the continuity of the intervention. At the end of the sixth month, the fourth home visit was paid, and after the final follow-up and measurements were performed, the patient was invited to the hospital and spirometry measurements were repeated. At the end of the study, carbon monoxide (CO) levels of the participants who stated that they quit smoking were measured and those with CO levels less than 5 ppm were accepted as non-smokers. This measurement was performed with a handheld carbon monoxide measuring device.

At the control group; No home visits were paid to the participants in the control group, they were invited to the hospital and were interviewed using the face-to-face interview method twice at the end of the first and sixth months, and measurements were performed. The researcher also given at the end of the sixth month, all of the nursing interventions, given to the intervention group, for the control group.

Intervention Education Material;The booklet prepared by the researcher based on the relevant literature. Then it took its final form after expert opinion was received and was published. In the booklet, information on the function of the lungs, the definition of COPD, symptoms of and factors causing COPD, relationship between the disease and smoking and effects of smoking cessation on COPD is given.

TTM-based Smoking Cessation Guide; The guide was prepared considering the needs of individuals at each stage according to the transtheoretical model. The guide introduces the characteristics of each stage of change of the model and shows what should be done to initiate the change in the individual, and information and strategies related to the issue. In the use of the guide, first the stage of change is determined using the Stages of Change Scale and then the procedure to be followed according to the guide is determined.

The nursing intervention performed in the present study involved home visits and six-month periodic follow-up, health education, smoking cessation intervention in line with motivational interviewing principles and telephone counseling processes.

Reminders; Between the third and fourth home visits, the participants were contacted through telephone calls once a month to ensure the continuity of the motivation and thus the continuity of the intervention

Sample size calculation; The sample size was determined using the Win episcope 2.0 program. The sample size was calculated as 78 with a 5% margin of error and at a 15% prevalence rate and 95% confidence interval, and it was decided to include 40 patients in the intervention group and 40 patients in the control group. However, due to the difficulties which arose in the data collection process, the planned number of people could not be reached. Therefore, after the completion of the pre-test measurements, the sample power was re-calculated using the G-Power Data Analysis program and the sample size was considered adequate (0.56-1.21). Then upon the completion of the data collection, the post-hoc power analysis (0.42-0.99) was performed. The study was completed including 68 people in the sample (33 in the intervention group and 35 in the control group).

Study budget;This research received no specific grant from any funding agency in the public, commercial, or not-for-profit sectors

Data analyses; Data were analyzed using the IBM SPSS V23. While the independent samples t-test and Mann Whitney U test were used to compare the intergroup data, the paired samples t-test and Wilcoxon test were used to compare intragroup pre-test and post-test values, and the chi-square test and Fisher Exact test were used to analyze the categorical data. p-values less than 0.05 were considered statistically significant. The Fisher Exact test was used to check the significance.

Ethical aspects; Study approval was given by The Ethics Committee of Non-invasive Researches (decision number:B.30.2.ODM.0.20.08/1184). All participants were informed about this study and obtained oral-written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being diagnosed with COPD
* Being >40 years old
* Being a smoker currently
* Not having a physical or mental problem preventing the person from filling in the questionnaires to be used in the study and from using telephone
* Using a mobile phone that is available at all times
* Living in the city center of Samsun, a city on the north coast of Turkey
* Not receiving any smoking cessation treatment at the time of the study
* Not having medical contraindication preventing spirometric evaluation

Exclusion Criteria:

* Patients with exacerbations in the last two months
* Having receiving smoking cessation treatment

Exclusion Criteria for those already included in the study;

* Not completing the home visits process
* Agreeing to participate in the study but then withdrawing from the study for any reason
* Being diagnosed with lung cancer

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Fagerström Test for Nicotine Dependence | 6 mounth
  The test developed by Fagerström, Heatherton and Kozlowski in 1992 includes 6 items each of which is rated on a different scale. A total score ranging from 0 to 4 indicates low nicotine dependence, from 5 to 6 indicates moderate dependence and from 7 to 10 indicates high independence. It was adapted by Uysal et al. (2004). Cronbach's alpha value was 0.79 in the present study.
Stages of Change (SOC) scale | 6 mounth
  Prochaska and Diclemente (1983) explained smoking cessation through the gradual change process and developed the questions of change. Accordingly, people select one of the following corresponding to his/her situation: Precontemplation: I do not consider quitting smoking in the next six months. Contemplation: I am planning to quit smoking in the next six months. Preparation: I am planning to quit in the next 30 days. Action: I quit smoking less than six months ago. Maintenance: I have not been smoking for more than six months.
Processes of Change (POC) scale | 6 mounth
  The scale developed by Prochaska et al. (1988) includes 30 items questioning the cognitive processes (15 items) and behavioral processes (15 items). Each process contains five sub-dimensions. It is a five-point Likert type scale. The options determine which methods an individual uses in behavior change. In the present study, Cronbach's Alpha values ranged between 0.61 and 0.92.
Self-Efficacy (SE) scale | 6 mounth
  The scale developed by Velicer et al. (1990) measures the degree of confidence an individual has in maintaining non-smoking behavior in situations triggering smoking. It was adapted by Koyun, Bodur and Eroğlu (2015). Cronbach's alpha values of was 0.93 in the present study. The scale consists of eight items rated on a 5-point Likert type scale. The lowest and highest possible scores to be obtained from the scale are 8 and 40 respectively. The higher the score is the more successful the person is.
Decisional Balance (DB) scale | 6 mounth
  The scale developed by Velicer et al. (1985) has 12 items in two sub-dimensions: Pros of change (6 items) and Cons of change (6 items). The Cronbach's Alpha value was 0.71 and 0.85 in the present study. The items of the scale are rated on a five-point likert type scale. The minimum and maximum possible scores to be obtained from the scale are 6 and 30 respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Figen Cavusoglu, Asst. Prof, Principal Investigator — Ondokuz Mayıs University; Ayse Beser, Prof, Study Director — Koç University; Oguz Kılınc, Prof, Study Chair — Dokuz Eylul University; Nazmiye Tibel Tuna, Asst Prof, Study Chair — Ondokuz Mayıs University

IPD SHARING:
Plan to Share IPD: No